CLINICAL TRIAL: NCT03956316
Title: Short-Term Outcomes of Total Shoulder Arthroplasty Using the Titan Modular Total Shoulder System
Status: Completed | Type: Observational
Sponsor: OrthoIndy (Other)
Collaborators: Integra LifeSciences Corporation (Industry)
Responsible Party: Principal Investigator, Troy Roberson, MD, Principal Investigator, OrthoIndy
Other Study IDs: Integra TSA
Record Dates: First submitted 2019-04-10; First posted 2019-05-20 (Actual); Last update posted 2019-05-20 (Actual); Status verified 2019-05

CONDITIONS: Shoulder Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

INTERVENTIONS:
Device: Titan Modular Total Shoulder System — total shoulder arthroplasty using the Titan Modular Total Shoulder System

SUMMARY:
The goals of total, reverse total and hemi shoulder arthroplasty are the same, to alleviate the patient's pain and obtain a full functional recovery. This outcome depends on the surgeon's ability to reproduce normal glenohumeral anatomy including bone morphology, capsular tension and rotator cuff function. Shoulder arthroplasty has become a safe and effective treatment for various diseases of the shoulder. This study goal is to document and report the short-term functional, radiographic, and quality of life outcomes of total shoulder arthroplasty (TSA) using the titan modular shoulder system.

ELIGIBILITY:
Inclusion Criteria:

* Total shoulder arthroplasty using the Titan Modular Total Shoulder System

Exclusion Criteria:

* Declining to participate

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 39 subjects received total shoulder arthroplasty using the Titan Modular Total Shoulder System. 25 subjects agreed to participate in the study.
Sampling Method: Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2014-10-15 (Actual); Primary Completion 2015-12-22 (Actual); Study Completion 2015-12-22 (Actual)

PRIMARY OUTCOMES:
ASES | two year post op
  1. ASES: the American Shoulder and Elbow Surgeons Standardized Shoulder Assessment
  1. The ASES scale is intended to measure functional limitations and pain of the shoulder.
  2. ASES is a 0 - 100 point scale; higher scores indicate better outcomes.
  i. The ASES consists of two dimensions: pain and function (worth 50 points each).
  a. The ASES questionnaire is composed of both a physician-rated component and a patient-reported component. Patient questions focus on: joint pain, instability and activities of daily living. Physician questions focus on: range of motion, strength, signs and instability
EQ-5D-5L | two year post op
  2. EQ5D-5L: EuroQuol-5D
  a. The EQ5D-5L scale evaluates general health status. The EQ-5D-5L has two sections; the first section measures health status using a descriptive system (index of 5 scores) and the second section measures health status on a Visual Analog Scale.
  i. The EQ-5D-5L VAS outcome is measured on a 0 - 100 point scale. Optimal health status is indicated with a score of 100.
  ii. The EQ-5D-5L descriptive system consists of 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension is evaluated with a score of 1-5, higher scores indicate worse outcomes.
  1. On each dimension, a score of 1 indicates no patient problems in that dimension, 2 indicates slight problems in that dimension, 3 indicates moderate problems in that dimension, 4 indicates severe problems in that dimension and 5 indicates extreme problems in that dimension.
PENN | two year post op
  3. PENN: PENN Shoulder Score
  1. The PENN Shoulder Score is used to assess patient self-reported levels of pain, satisfaction and function.
  2. PENN is measured on a 0 - 100 point scale; higher scores indicate better outcomes.
  3. The PENN consists of 3 subscales: pain (at rest, with activity, and with strenuous activity), satisfaction and function. The PENN Pain subscale is scored from 0 to 30, the PENN satisfaction subscale is scored from 0 to 10 and the PENN function subscale is scored from 0 to 60.
SANE | two year post op
  4. SANE: Single assessment numeric evaluation
  1. SANE is an outcome scale used to record the patient's self-reported function.
  2. SANE is implemented on a scale of 0 - 100, 100 indicates full function (or function prior to injury) and 0 represents no function.
CS | two year post op
  5. CS: Constant-Murley Score
  1. The CS score assesses functionality after the treatment of a shoulder injury.
  2. CS is measured on a 0 - 100 point scale. Higher scores indicate better shoulder function.
  3. CS is composed of four subscales: pain (15 points, based on patient report), activities of daily living (20 points, based on patient report), strength (25 points), and range of motion (40 points).
WOOS | two year post op
  6. WOOS: Western Ontario Osteoarthritis of the Shoulder index
  1. WOOS is a disease-specific quality of life PRO tool, developed for osteoarthritis.
  2. WOOS is measured on a 0-1900 point scale; 1900 indicates a clinical outcome fully symptomatic of osteoarthritis and 0 indicates an asymptomatic outcome.
  i. WOOS is composed of 19 items scored on 100-point VAS scales. The 19 items represent four domains (6 questions for pain and physical symptoms, 5 questions for sport/recreation/work function, 5 questions for lifestyle function and 3 questions for emotional function).

IPD SHARING:
Plan to Share IPD: No
Data will not be shared.